CLINICAL TRIAL: NCT03038945
Title: Barbed vs Standard Suture for Laparoscopic Vaginal Cuff Closure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CES University (Other)
Responsible Party: Principal Investigator, Claudia López, Gynecologist, CES University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 377
Record Dates: First submitted 2017-01-19; First posted 2017-02-01 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Gynecologic Surgical Procedures
Keywords: Laparoscopy; Hysterectomy; Suture Techniques

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2/0 barbed suture (Experimental): Use barbed suture for the closure of the vaginal vault in patients with total Laparoscopic hysterectomy caused by a benign gynecologist pathology
  Interventions: Other: 2/0 barbed suture
- Vicryl suture (Active Comparator): Use VICRYL suture for the closure of the vaginal vault in patients with total Laparoscopic hysterectomy caused by a benign gynecologist pathology
  Interventions: Other: 0/0 Vicryl suture

INTERVENTIONS:
Other: 2/0 barbed suture — Close vaginal vault 2 planes with 2/0 barbed suture in patients with total laparoscopic hysterectomy in benign pathology
  Arms: 2/0 barbed suture
Other: 0/0 Vicryl suture — Close vaginal vault 2 planes with 0/0 Vicryl suture in patients with total laparoscopic hysterectomy in benign pathology
  Arms: Vicryl suture

SUMMARY:
Total laparoscopic hysterectomy is a procedure that is performed each time more often. One of the problems described for this procedure has to do with the closure of the vaginal vault, increased surgical time when suture laparoscopically, complications such as dehiscence of the dome, infections, hematomas and dyspareunia. A prospective study will be conducted to compare two different techniques for closure of the vaginal vault.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for total laparoscopic hysterectomy without other simultaneous procedures , for benign causes , who were agree to participate in the trial and give their written consent.
* Patients ASA (American Society of Anesthesiologists) 1 and 2
* Patients who are able to communicate by telephone and answer questions

Exclusion Criteria:

* Patients with coagulation disorders, chronic use of corticosteroids, COPD (chronic obstructive pulmonary disease), collagen diseases, diabetes.
* Endometriosis III / IV
* Patients who can not be reached by phone

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2016-10; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Cuff closure time | 20 minutes
  time spend for vaginal Cuff closure (in minutes)

SECONDARY OUTCOMES:
Intra or postoperative complications | 10 days
  Clinical follow-up to complications during the surgery and ten days after, through questions and clinical exam.
Dyspareunia | 12 weeks
  the visual scale was used to analyze the dyspareunia

CONTACTS AND LOCATIONS:
Overall Officials: CLAUDIA LOPEZ, Gynecologist, Principal Investigator — CLINICA DEL PRADO
Locations (1):
- Claudia Lopez, Medellín, Antioquia, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cohen SL, Einarsson JI. Total and supracervical hysterectomy. Obstet Gynecol Clin North Am. 2011 Dec;38(4):651-61. doi: 10.1016/j.ogc.2011.09.002. PMID 22134014
- [Result] Hur HC, Donnellan N, Mansuria S, Barber RE, Guido R, Lee T. Vaginal cuff dehiscence after different modes of hysterectomy. Obstet Gynecol. 2011 Oct;118(4):794-801. doi: 10.1097/AOG.0b013e31822f1c92. PMID 21934442
- [Result] Ceccaroni M, Berretta R, Malzoni M, Scioscia M, Roviglione G, Spagnolo E, Rolla M, Farina A, Malzoni C, De Iaco P, Minelli L, Bovicelli L. Vaginal cuff dehiscence after hysterectomy: a multicenter retrospective study. Eur J Obstet Gynecol Reprod Biol. 2011 Oct;158(2):308-13. doi: 10.1016/j.ejogrb.2011.05.013. Epub 2011 Jul 1. PMID 21723030
- [Result] Einarsson JI, Vellinga TT, Twijnstra AR, Chavan NR, Suzuki Y, Greenberg JA. Bidirectional barbed suture: an evaluation of safety and clinical outcomes. JSLS. 2010 Jul-Sep;14(3):381-5. doi: 10.4293/108680810X12924466007566. PMID 21333192
- [Result] Hwang JH, Lee JK, Lee NW, Lee KW. Vaginal cuff closure: a comparison between the vaginal route and laparoscopic suture in patients undergoing total laparoscopic hysterectomy. Gynecol Obstet Invest. 2011;71(3):163-9. doi: 10.1159/000316052. Epub 2010 Dec 14. PMID 21160140
- [Result] Jeung IC, Baek JM, Park EK, Lee HN, Kim CJ, Park TC, Lee YS. A prospective comparison of vaginal stump suturing techniques during total laparoscopic hysterectomy. Arch Gynecol Obstet. 2010 Dec;282(6):631-8. doi: 10.1007/s00404-009-1300-0. Epub 2009 Nov 27. PMID 19943055
- [Result] Siedhoff MT, Yunker AC, Steege JF. Decreased incidence of vaginal cuff dehiscence after laparoscopic closure with bidirectional barbed suture. J Minim Invasive Gynecol. 2011 Mar-Apr;18(2):218-23. doi: 10.1016/j.jmig.2011.01.002. PMID 21354068
- [Result] Uccella S, Ghezzi F, Mariani A, Cromi A, Bogani G, Serati M, Bolis P. Vaginal cuff closure after minimally invasive hysterectomy: our experience and systematic review of the literature. Am J Obstet Gynecol. 2011 Aug;205(2):119.e1-12. doi: 10.1016/j.ajog.2011.03.024. Epub 2011 Mar 22. PMID 21620360
- [Result] Ramirez PT, Klemer DP. Vaginal evisceration after hysterectomy: a literature review. Obstet Gynecol Surv. 2002 Jul;57(7):462-7. doi: 10.1097/00006254-200207000-00023. PMID 12172223
- [Result] Iaco PD, Ceccaroni M, Alboni C, Roset B, Sansovini M, D'Alessandro L, Pignotti E, Aloysio DD. Transvaginal evisceration after hysterectomy: is vaginal cuff closure associated with a reduced risk? Eur J Obstet Gynecol Reprod Biol. 2006 Mar 1;125(1):134-8. doi: 10.1016/j.ejogrb.2005.08.009. Epub 2005 Sep 8. PMID 16154253
- [Result] Croak AJ, Gebhart JB, Klingele CJ, Schroeder G, Lee RA, Podratz KC. Characteristics of patients with vaginal rupture and evisceration. Obstet Gynecol. 2004 Mar;103(3):572-6. doi: 10.1097/01.AOG.0000115507.26155.45. PMID 14990423
- [Result] Jacoby VL, Autry A, Jacobson G, Domush R, Nakagawa S, Jacoby A. Nationwide use of laparoscopic hysterectomy compared with abdominal and vaginal approaches. Obstet Gynecol. 2009 Nov;114(5):1041-1048. doi: 10.1097/AOG.0b013e3181b9d222. PMID 20168105
- [Result] Cronin B, Sung VW, Matteson KA. Vaginal cuff dehiscence: risk factors and management. Am J Obstet Gynecol. 2012 Apr;206(4):284-8. doi: 10.1016/j.ajog.2011.08.026. Epub 2011 Aug 27. PMID 21974989
- [Result] Uccella S, Ceccaroni M, Cromi A, Malzoni M, Berretta R, De Iaco P, Roviglione G, Bogani G, Minelli L, Ghezzi F. Vaginal cuff dehiscence in a series of 12,398 hysterectomies: effect of different types of colpotomy and vaginal closure. Obstet Gynecol. 2012 Sep;120(3):516-23. doi: 10.1097/AOG.0b013e318264f848. PMID 22914459
- [Result] Chan WS, Kong KK, Nikam YA, Merkur H. Vaginal vault dehiscence after laparoscopic hysterectomy over a nine-year period at Sydney West Advanced Pelvic Surgery Unit - our experiences and current understanding of vaginal vault dehiscence. Aust N Z J Obstet Gynaecol. 2012 Apr;52(2):121-7. doi: 10.1111/j.1479-828X.2012.01411.x. Epub 2012 Feb 15. PMID 22335453
- [Result] Blikkendaal MD, Twijnstra AR, Pacquee SC, Rhemrev JP, Smeets MJ, de Kroon CD, Jansen FW. Vaginal cuff dehiscence in laparoscopic hysterectomy: influence of various suturing methods of the vaginal vault. Gynecol Surg. 2012 Nov;9(4):393-400. doi: 10.1007/s10397-012-0745-5. Epub 2012 May 3. PMID 23144640
- [Result] ACOG Committee Opinion No. 444: choosing the route of hysterectomy for benign disease. Obstet Gynecol. 2009 Nov;114(5):1156-1158. doi: 10.1097/AOG.0b013e3181c33c72. PMID 20168127
- [Result] Hur HC, Guido RS, Mansuria SM, Hacker MR, Sanfilippo JS, Lee TT. Incidence and patient characteristics of vaginal cuff dehiscence after different modes of hysterectomies. J Minim Invasive Gynecol. 2007 May-Jun;14(3):311-7. doi: 10.1016/j.jmig.2006.11.005. PMID 17478361
- [Result] Kho RM, Akl MN, Cornella JL, Magtibay PM, Wechter ME, Magrina JF. Incidence and characteristics of patients with vaginal cuff dehiscence after robotic procedures. Obstet Gynecol. 2009 Aug;114(2 Pt 1):231-235. doi: 10.1097/AOG.0b013e3181af36e3. PMID 19622982
- [Result] Villa MT, White LE, Alam M, Yoo SS, Walton RL. Barbed sutures: a review of the literature. Plast Reconstr Surg. 2008 Mar;121(3):102e-108e. doi: 10.1097/01.prs.0000299452.24743.65. PMID 18317092
- [Result] Greenberg JA. The use of barbed sutures in obstetrics and gynecology. Rev Obstet Gynecol. 2010 Summer;3(3):82-91. PMID 21364859